CLINICAL TRIAL: NCT02709252
Title: Effect of the Pneumoperitoneum on Dynamic Variables Delta PP and PVI During Trendelenburg Position.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Forget Patrice, PI, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201134
Record Dates: First submitted 2016-03-03; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Surgery

ARMS (1):
- Cohort (Experimental): Only one cohort is included with comparisons of two different hemodynamic parameters
  Interventions: Device: PVI and deltaPP after trendelenburg position change

INTERVENTIONS:
Device: PVI and deltaPP after trendelenburg position change — Comparison of hemodynamic parameters during surgery after position change

SUMMARY:
Arterial pulse pressure variation induced by mechanical ventilation (ΔPP) is considered one of the best parameter to predict fluid responsiveness in patients under general anaesthesia. Pleth Variability Index (PVI) has been proposed as a less invasive alternative. However, the pneumoperitoneum has been recently seen suggested as a limitation to their interpretation. The aim of this observational study is to compare changes in ΔPP and PVI related to autotransfusion associated with a Trendelenburg manoeuver before and during laparoscopy in patients undergoing elective surgery.

ELIGIBILITY:
* American Society of Anesthesiologists (ASA) score I-II
* scheduled for elective abdominal laparoscopic surgery
* with written informed consent
* more than 18 years
* Body Mass Index < 40 kg.m-2
* no supraventricular arrhythmias
* no heart failure with ejection fraction <25 %
* no peripheral vascular
* no severe respiratory disease
* no end stage renal failure (creatinine clearance <30ml/min).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pleth variability index (in %) | 5 minutes
  Before/after trendelenburg positioning in laparoscopic surgery
Pulse Pressure variation (deltaPP) (in %) | 5 minutes
  Before/after trendelenburg positioning in laparoscopic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Brugmann hospital, Brussels, Belgium